CLINICAL TRIAL: NCT04979000
Title: The Role of High-risk HPV in Sinonasal Carcinomas: a Retrospective Tissue Analysis of the Increasing Frequency and Case-control Study to Evaluate the Association of HPV Serology and Behavioral Risk Factors
Brief Title: HPV in Sinonasal Ca: Retrospective Analysis Association of Human Papilloma Virus (HPV) Serology and Behavioral Risk Factors
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: J20108; IRB00270617 (Other: JHM IRB)
Record Dates: First submitted 2021-07-09; First posted 2021-07-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Sinonasal Carcinoma; HPV-Related Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For cases, paraffin embedded tumor samples will be tested for HPV. The blood sample collected at baseline (both cases and controls) will be tested for HPV antibodies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with a confirmed diagnosis of sinonasal cancer.
- Controls: Patients being seen for benign conditions at Johns Hopkins.

SUMMARY:
This is a case-control study designed to evaluate the role of anatomic site, gender and race in human papillomavirus-associated head and neck squamous cell cancers (HNSCC). We will explore the role of HPV, tobacco, alcohol and drug use, in HNSCC by tumor site with particular emphasis on the sinonasal cavity as well as differences in risk factors for HPV-positive HNSCC by gender and race.

ELIGIBILITY:
Inclusion Criteria:

* Cases:

  * Patients must be 18 years of age or older with a confirmed or suspected diagnosis of sinonasal cancer
  * Patients must have either a routine diagnostic biopsy of primary tumor or surgical resection planned as part of routine care (to allow for the collection of tumor sample for the study) or grant access to archival material, from a previously performed biopsy.
  * Willing to provide 20 mL blood sample
  * Ability to understand and the willingness to sign a written informed consent document
* Controls:

  * Must be 18 years of age or older within the categories of age, gender, and race needed to match cases
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Cases:

  * Presence of medical or psychiatric condition affecting ability to give voluntary, informed consent
  * Participants who do not speak English and do not agree to use of a telephone or video interpreter will be excluded. However, if there is a hearing, literally or minor fluency issue and the participant requests assistance from a family member or the study coordinator, this individual may still enroll and receive this assistance to ensure they fully hear and understand everything being asked
* Controls:

  * Presence of medical or psychiatric condition affecting ability to give voluntary, informed consent
  * Participants who do not speak English and do not agree to use of a telephone or video interpreter will be excluded. However, if there is a hearing, literacy or minor fluency issue and the participant requests assistance from a family member or the study coordinator, this individual may still enroll and receive this assistance to ensure they fully hear and understand everything being asked
  * No prior diagnosis of head and neck cancer, except basal cell cancer
  * No previous radiation therapy of the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases:
  Patients with a confirmed diagnosis of sinonasal cancer, or clinical findings consistent with this diagnosis, seen in the Departments of Otolaryngology/Head and Neck Surgery, Radiation Oncology, or Medical Oncology of the Johns Hopkins Sidney Kimmel Comprehensive Cancer Center (SKCCC) or Johns Hopkins Head and Neck Surgery at Suburban Hospital are eligible for this study.
  Controls:
  Patients seen for benign conditions in the same Departments of Otolaryngology/Head and Neck Surgery, Radiation Oncology, and Medical Oncology at SKCCC or Suburban Hospital are eligible for enrollment as non-cancer controls in this study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
HPV Status | Collected at time of surgery or previously conducted biopsy
  High risk HPV present or absent in tumor

SECONDARY OUTCOMES:
Gender Differences | completion of the study, approximately 2 years
  Gender differences in HPV-HNSCC risk factors (tobacco, alcohol, drug use and sexual behavior).
Race/Ethnicity Differences | completion of the study, approximately 2 years
  Race/ethnicity differences in HPV-HNSCC risk factors (tobacco, alcohol, drug use and sexual behavior).

CONTACTS AND LOCATIONS:
Overall Officials: Nyall London, M.D., Principal Investigator — Department of Otolaryngology and Surgery
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States